CLINICAL TRIAL: NCT00332228
Title: Study Behavioral Naltrexone Therapy: A Novel Treatment for Heroin Dependence
Brief Title: Behavioral Naltrexone Therapy: A Novel Treatment for Heroin Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 5004-R; R01DA010746 (NIH)
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Opiate Dependence
Keywords: opiate dependence; heroin dependence; naltrexone; cognitive behavioral therapy
MeSH Terms: conditions — Opioid-Related Disorders; Heroin Dependence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CE plus oral +depot naltrexone (Active Comparator): Compliance enhancement (CE), simulating standard treatment with oral naltrexone plus two depot naltrexone;
  Interventions: Drug: depot naltrexone; Behavioral: Compliance enhancement (CE)
- CE plus oral naltrexone+ placebo (Placebo Comparator): CE with oral naltrexone plus two placebo injections
  Interventions: Behavioral: Compliance enhancement (CE)
- BNT plus Depot naltrexone (Experimental): BNT plus two doses of depot naltrexone prior to hospital discharge
  Interventions: Drug: depot naltrexone; Drug: BNT
- BNT plus PBO injection (Placebo Comparator): BNT plus two placebo injections
  Interventions: Drug: BNT

INTERVENTIONS:
Drug: depot naltrexone — long-acting depot parenteral formulation of naltrexone
  Arms: BNT plus Depot naltrexone; CE plus oral +depot naltrexone
Behavioral: Compliance enhancement (CE) — Compliance enhancement (CE), simulating standard treatment with oral naltrexone
  Arms: CE plus oral +depot naltrexone; CE plus oral naltrexone+ placebo
Drug: BNT — behavioral therapy with oral naltrexone maintenance for the treatment of heroin addiction
  Arms: BNT plus Depot naltrexone; BNT plus PBO injection

SUMMARY:
The overall goal of this research project is to test the efficacy of a newly developed therapy, Behavioral Naltrexone Therapy (BNT), to enhance the success of naltrexone maintenance and long-term abstinence for individuals with heroin dependence. This study includes free detox and outpatient treatment for opioid dependence that includes medication and a behavioral intervention.

DETAILED DESCRIPTION:
The goal of this Stage II project is to test the efficacy of a new combination of behavioral therapy with oral naltrexone maintenance for the treatment of heroin addiction, and to test a new long-acting depot parenteral formulation of naltrexone in initiating treatment.

1. Outpatient treatment with Behavioral Naltrexone Therapy will yield a lower rate of relapse to illicit opiates compared to naltrexone plus compliance enhancement therapy. Hypotheses:
2. Injections of depot naltrexone will reduce early attrition, improve initial stabilization on oral naltrexone, and improve long-term outcome, particularly when combined with Behavioral Naltrexone Therapy.
3. Patients who exhibit escalating levels of commitment language strength throughout one early session of BNT will remain in treatment longer, will take more doses of naltrexone, and will provide a higher percentage of opiate-free urines.
4. Increased commitment language strength on the part of the SO monitor will contribute independently to the outcome of the identified patient, when controlling for patient level commitment.

A critical objective of this current proposal is to improve retention, particularly in the initial weeks of treatment. Preliminary work with a new depot formulation of naltrexone was conducted (Comer et al, 1999, unpublished data), showing that it is well tolerated and provides therapeutic blood levels and blockade of opiate effects for up to four weeks after a single injection. By removing the option of stopping naltrexone to sample heroin, a common mode of relapse, we hope to prevent early attrition and fully expose all patients to the behavioral regimen of BNT, intended to shape strong compliance with oral naltrexone and motivation for abstinence and lifestyle change.

160 heroin-dependent individuals seeking treatment will be recruited at PI (STARS) or referred from other sites (e.g., private physician; other detoxification programs). Prospective patients will be offered hospitalization for detoxification for rapid transition to naltrexone followed by outpatient naltrexone maintenance and counseling for six months. All enrolled participants will be encouraged to return for follow-up assessment visits at one, three, and six months beyond the completion of their participation for research purposes.

Patients will be randomly assigned to either the newly developed BNT or Compliance Enhancement Therapy (CET), a manual-guided approach developed by Carroll and O'Malley at Yale University as a control condition for psychotherapy studies with substance dependent patients. Patients will also be randomly assigned to receive either active or placebo injections of depot naltrexone prior to discharge from the detoxification. Therefore, there will be four treatment conditions with 40 participants per condition. These four conditions include: 1) BNT plus two doses of depot naltrexone prior to hospital discharge; 2) BNT plus two placebo injections; 3) Compliance Enhancement (CE), simulating standard treatment with oral naltrexone plus two depot naltrexone injections; and 4) CE plus two placebo injections.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, aged 18-60. Clinical Interview.
2. Meets DSM-IV criteria for current opiate dependence disorder, supported by a positive urine for opiates and a positive naloxone challenge test if the diagnosis is unclear. If participating as an outpatient only, recent opiate dependence must be confirmed by clinical history and/or communication with former treatment provider.

   Clinical and SCID interview. Urine toxicology. Naloxone Challenge (see Procedures) Communication with former treatment provider.
3. Able to give informed consent. Clinical interview and mental status exam
4. There must be one qualified significant other who is willing to be interviewed and participate in program in order for a subject to be included in the study.

Clinical interview, and statement by significant other.

Exclusion Criteria:

1. Pregnancy, lactation, or failure in a sexually active woman to use adequate contraceptive methods.

   Clinical Interview, physical examination, serum pregnancy test
2. Active medical illness which might make participation hazardous, such as untreated hypertension, acute hepatitis with SGOT or SGPT levels >2-3 times normal, unstable diabetes, chronic organic mental disorder (e.g., AIDS dementia).

   Clinical Interview, physical examination, laboratory (Chem-20, CBC, urinalysis), ECG
3. Active psychiatric disorder which might interfere with participation or make participation hazardous, including DSM-IV schizophrenia, bipolar disorder with mania or psychosis, and depressive disorder with suicide risk or 1 or more suicide attempts within the past year.

   Clinical and SCID interview, clinical mental status examination, discussions with previous psychiatrist or treatment provider if formerly in treatment.
4. History of allergic reaction to buprenorphine, naloxone, naltrexone, clonidine, or clonazepam.

   Clinical Interview
5. Currently prescribed or regularly taking opiates for chronic pain or medical illness.

   Clinical Interview
6. Current participation in another intensive substance abuse treatment program.

   Clinical Interview
7. Current participation in a methadone maintenance treatment program and/or regular use of illicit methadone (>30 mg per week). Clinical Interview; Urine toxicology.
8. Only available significant other is an active substance abuser, has an active psychiatric or medical illness which would interfere with participation (e.g., chronic psychosis, depression with suicide risk), or has a history of significant physical violence with the participant.

   Clinical Interview
9. History of accidental drug overdose in the last three years as defined as an episode of opioid-induced unconsciousness or incapacitation, whether or not medical treatment was sought or received.

Clinical Interview

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2002-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
proportion of patients relapsing to illicit opiates based on urine toxicology and self report. | over 6 months of trial or length of participation
  proportion of patients relapsing to opiate use
proportion of patients retained in treatment | over course of 6 months of trial
  proportion of patients retained over the course of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Edward Nunes, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - New York State Psychiatric Institute, New York, New York
  - STARS, New York, New York

REFERENCES:
- See also: serive website — http://www.stars.columbia.edu